CLINICAL TRIAL: NCT02732366
Title: Living in Fitness Together (LIFT): Testing an Innovative Fall Prevention Program
Acronym: LIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Mt. Ascutney Hospital and Health Center (Other); Foundation for Physical Therapy, Inc. (Industry); Boston University (Other)
Responsible Party: Principal Investigator, Christine McDonough, Assistant Professor of Physical Therapy, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO18020039
Record Dates: First submitted 2016-03-24; First posted 2016-04-08 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Accidental Falls
Keywords: aged [MeSH term]; exercise [MeSH term]

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-based exercise and peer coaching (Experimental): This treatment arm will include physical therapist-led group-based exercise, goal-setting, peer coaching training, individualized home program, and activity monitoring.
  Interventions: Behavioral: Group-based exercise and peer coaching
- Usual PT and attention control grp class (Active Comparator): This arm consists of the continuation of one-on-one PT along with participation in an attention control - healthy living class.
  Interventions: Other: Usual PT and attention control grp class

INTERVENTIONS:
Behavioral: Group-based exercise and peer coaching — Group-based exercise and peer coaching will take place over 6 weeks plus one booster visit after 3 months, and include physical therapist-led 1 hour sessions 2 times per week for 2 weeks followed by once per week for 4 weeks (8 sessions) to include: progressive strengthening, balance and mobility exercises; patient goal setting; peer coaching training activities to teach group members ways to help each other to meet their exercise goals during and after classes are over. There will be an individualized home program including flexibility, strengthening, walking, and balance, as well as activity monitoring.
  Arms: Group-based exercise and peer coaching
Other: Usual PT and attention control grp class — The usual PT and attention control group class will receive standard one-on-one PT strength, balance, gait and education intervention, and group classes to provide valuable information about healthy living, including nutrition, relaxation, and stress management. The attention control - healthy living group classes will take place over 6 weeks plus one booster visit after 3 months, and include 1 hour sessions 2 times per week for 2 weeks followed by once per week for 4 weeks (8 sessions).
  Arms: Usual PT and attention control grp class

SUMMARY:
The purpose of this study is to test the feasibility and preliminary efficacy of a group-based fall prevention program for older adults.

DETAILED DESCRIPTION:
Falls are the leading cause of non-fatal and fatal injuries in older adults. The number of fall-related older adult deaths in 2005 reached 15,802. Overall, thirty percent of adults over the age of 65 fall every year, and the risk for falls increases dramatically with age. Direct medical costs related to falls reached $19 billion in 2000. In 2006 a national study found that 5.8 million older adults (16%) reported a fall in the prior 3 month period and 1.8 million had been injured. Falls and fall-related injuries have an important impact on mobility, functioning, and the quality of life of older adults, and for many, result in catastrophic mobility decline, loss of independence and institutionalization. The trends in falls and aging in the population make this a critical problem for our time.

Current evidence and guidelines recommend assessment of several important risk factors and providing individualized intervention for older adults at increased risk of falls. Strength, balance and gait training are among the most potent intervention elements. Evidence shows that fall risk benefits gained from exercise are completely lost within 12 weeks if exercise is not continued. Therefore, persistence with exercise and physical activity are critical to the long-term success of fall prevention treatments. The proposed project tests the feasibility and preliminary efficacy of an innovative group-based fall prevention program called Living In Fitness Together (LIFT). The program consists of group-based physical therapy for strength, balance, mobility and flexibility training, an individualized home program including walking for physical activity, and training of the group members to support and coach each other toward meeting their exercise and physical activity goals. It consists of 8 group sessions over 6 weeks plus one group booster session delivered by a physical therapist, occupational therapist and trained staff. The program is designed to deliver progressive, tailored, and challenging exercise intervention for older adults at risk for falls and empower older adults to meet their goals for exercise and physical activity through training in self-management, and peer-coaching within the exercise group. The aim of this project is to test the feasibility of implementing the fall prevention program with peer-coaching in the context of physical therapy practice, and to assess its safety and initial efficacy. The results of this study will be the foundation of a formal clinical trial of a novel program of exercise and peer- coaching for exercise adherence. This program has potential to be incorporated into physical therapy practice and disseminated widely, and to have an important impact on the number of falls and fall-related injuries that occur in older adults.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 65 and over
* at risk for falls as identified by health care provider
* able to participate in group exercise with upper extremity support for balance (e.g. chair)

Exclusion Criteria:

* active vertigo, postural hypotension, unstable cardiac conditions
* major neurological disorders such as Parkinson's disease, recent major cerebrovascular event, multiple sclerosis, amyotrophic lateral sclerosis

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M McDonough, PT, MS, PhD, Principal Investigator — University of Pittsburgh, School of Health and Rehabilitation Sciences, Department of Physical Therapy
Locations (1):
- Mount Ascutney Hospital and Health Center, Windsor, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stevens JA, Corso PS, Finkelstein EA, Miller TR. The costs of fatal and non-fatal falls among older adults. Inj Prev. 2006 Oct;12(5):290-5. doi: 10.1136/ip.2005.011015. PMID 17018668
- [Background] Moyer VA; U.S. Preventive Services Task Force. Prevention of falls in community-dwelling older adults: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2012 Aug 7;157(3):197-204. doi: 10.7326/0003-4819-157-3-201208070-00462. PMID 22868837
- See also: Fatalities and injuries from falls among older adults - US 1993-2003 and 2001-2005. Morbidity and mortality weekly report. 2006 — http://www.cdc.gov/mmwr/preview/mmwrhtml/mm5545a1.htm
- See also: Self-reported falls and fall-related injuries among persons aged >65 years - US, 2006. Morbidity and mortality weekly report. 2008 — http://www.cdc.gov/mmwr/preview/mmwrhtml/mm5709a1.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from physician and physical therapist practices in a rural regional hospital. The intervention and control conditions were provided as 8-week programs. Recruitment was coordinated to occur approximately 4 weeks prior to a scheduled program/session, until sufficient numbers of participants were identified.
Pre-assignment Details: Two participants withdrew after consenting and before randomization. Note that randomization was done in session blocks.
Period: Overall Study
Arm/Group | Group-based Exercise and Peer Coaching | Usual PT and Attention Control Grp Class
Started | 23 | 23
Withdrawal by Participant | 5 | 2
Completed | 18 | 21
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Population: There were 7 withdrawals from the study between randomization and baseline testing/program start. Therefore the baseline analysis population is 39.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group-based Exercise and Peer Coaching | Usual PT and Attention Control Grp Class | Total
Number analyzed (Participants) | 18 | 21 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (5.6) | 77.2 (6.7) | 76.4 (6.17)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: missing: 1
  Participants
    number analyzed (Participants) | 18 | 20 | 38
    Female | 13 | 13 | 26
    Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 20 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 21 | 39
Timed Up and Go (seconds) [Mean (Standard Deviation); unit: seconds] — The Timed Up and Go is a physical performance measure that measures leg strength, mobility and fall risk using stopwatch, standard arm chair, and a line marked on the floor at 3 meters/10 feet away from the front edge of the chair. The participant may use walking aid and push off of the chair to stand up. The participant begins seated in the chair. When prompted with "Go" the participant stands, walk to the mark, turns, walks back an sits down. The results are reported in seconds.
  seconds | 12.6 (2.3) | 16.7 (9.0) | 14.65 (6.57)
30 Second Chair Stand [Mean (Standard Deviation); unit: number of stands] — This is a performance-based measure. The equipment needed includes a chair with a straight back without arm rests (seat 17 inches high) and a stopwatch. The participant sits in the chair, places hands on opposite shoulders crossed at the wrists with feet on the floor with back straight. On the verbal prompt "GO" the participant rises to a full standing position, sits back down, and repeats as many times as possible within 30 seconds. Age and gender-stratified thresholds have been established for fall risk.
  number of stands | 8.89 (3.5) | 8.24 (4.1) | 8.56 (3.74)

OUTCOME MEASURES:

1. Primary Outcome: Enrollment
Description: To assess feasibility of the intervention, the number of patients identified as eligible, the number who refuse to participate, and the number who enroll in the study will be collected.
Time Frame: 6 months
Population: 342 older adults were screened for eligibility.
Measure: Number; unit: participants
Groups:
- Screened Population: Number screened
Arm/Group | Screened Population
Number analyzed (Participants) | 342
participants
  Screened | 342
  Did not meet inclusion criteria | 142
  Met at least one exclusion criterion met | 23
  Eligible | 177
  Not interested | 101
  Unable to attend sessions | 25
  Could not be reached | 3
  Enrolled | 48

2. Primary Outcome: Intervention and Control Group Program Attendance
Description: To assess feasibility of the intervention, the percentage of sessions attended by patients enrolled in the study will be collected.
Time Frame: 6 weeks
Measure: Number; unit: percentage of sessions
Groups:
- Group-based Exercise and Peer Coaching: Attendance to 8 intervention sessions for 6 groups
- Usual PT and Attention Control Grp Class: Attendance to 6 control group sessions for 6 groups
Arm/Group | Group-based Exercise and Peer Coaching | Usual PT and Attention Control Grp Class
Number analyzed (Participants) | 18 | 21
percentage of sessions | 85.5 | 95.0

3. Primary Outcome: Program Completion
Description: To assess feasibility of the intervention, the number of patients who complete the program will be collected.
Time Frame: 6 weeks
Population: The number of participants that attended 6 week program (non-withdrawals).
Measure: Number; unit: number of participants
Arm/Group | Group-based Exercise and Peer Coaching | Usual PT and Attention Control Grp Class
Number analyzed (Participants) | 18 | 21
number of participants | 18 | 20

4. Primary Outcome: Adverse Events
Description: To assess safety of the intervention, patients will be instructed to report all adverse events to the clinical investigators.
Time Frame: 6 months
Population: Participants in the intervention and control groups
Measure: Count of Participants; unit: Participants
Arm/Group | Group-based Exercise and Peer Coaching | Usual PT and Attention Control Grp Class
Number analyzed (Participants) | 18 | 21
Participants
  Number of Participants with AEs | 10 | 10
  Number of Participants with falls | 10 | 9

5. Primary Outcome: Adverse Events - Number of Events
Description: Number of Adverse Events
Time Frame: 6 months
Population: Number of Adverse Events
Measure: Number; unit: number of events
Arm/Group | Group-based Exercise and Peer Coaching | Usual PT and Attention Control Grp Class
Number analyzed (Participants) | 18 | 21
number of events
  Falls | 14 | 13
  All non-fall adverse events | 1 | 4

ADVERSE EVENTS:
Time Frame: From baseline to 6 months from baseline
Description: Although falls were expected in this study, they were collected.
Arm/Group | Group-based Exercise and Peer Coaching | Usual PT and Attention Control Grp Class
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/18 | 2/21
Other Adverse Events (participants affected / at risk) | 10/18 | 10/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group-based Exercise and Peer Coaching (N=18) | Usual PT and Attention Control Grp Class (N=21)
heart attack (Cardiac disorders) | 0 (0) | 1 (1) — The participant reported having a heart attack during the follow-up period of the study, was treated in the hospital and by physician.
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) — the participant was admitted to the hospital for a urinary tract infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group-based Exercise and Peer Coaching (N=18) | Usual PT and Attention Control Grp Class (N=21)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — The participant experienced pneumonia and recovered.
spine disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Surgery for spinal stenosis
colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — experienced symptoms related to colitis
Falls (General disorders) | 10 (14) | 9 (13) — Falls
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) — urinary tract infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT02732366/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT02732366/ICF_001.pdf